CLINICAL TRIAL: NCT00882921
Title: A Multi-Center Observational Study Evaluating Anti-Idursulfase Serum Antibody Response in Hunter Syndrome Patients Enrolled in the Hunter Outcome Survey (HOS) Receiving Idursulfase Enzyme Replacement Therapy
Brief Title: An Observational Study Evaluating Anti-Idursulfase Serum Antibody Response in Hunter Syndrome Patients
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: HGT-ELA-042
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Results first posted 2014-07-30 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Hunter Syndrome
Keywords: MPS 2; MPSII; hunter's disease treatment; enzyme replacement therapy; hunter's disease; iduronate 2 sulfatase; mps diagnosis; mps symptoms; iduronate sulfatase; MPS II treatment; chronic ear infection; hunters syndrome; mps ii therapy; MPS2; hunter's syndrome; Hunter syndrome; elaprase; lysosomal storage disease; hunter syndrome therapy; mps society; hunter syndrome treatment; hunter's syndrome treatment; mucopolysaccharides; mps ii; idursulfase; hunters disease; enlarged adenoids; ert treatment; hunter disease; lysosomal storage disorder
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death; Lysosomal Storage Diseases | interventions — idursulfase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elaprase: Idursulfase 0.5 mg/kg Weekly
  Interventions: Biological: Idursulfase

INTERVENTIONS:
Biological: Idursulfase — Patients received idursulfase as prescribed by their physician following locally approved prescribing information. Patients will not be provided idursulfase by Shire Human Genetic Therapies, Inc. or the HOS.
  Other Names: Elaprase

SUMMARY:
The objective of this study is to evaluate the effect of anti-idursulfase antibodies on idursulfase safety (measured by infusion related adverse events) between patients who develop anti-idursulfase antibodies and patients who do not after long-term idursulfase enzyme replacement therapy (ERT).

DETAILED DESCRIPTION:
This study is being conducted to satisfy post-marketing commitments to monitor anti-idursulfase antibody development in Hunter syndrome patients after long-term idursulfase enzyme replacement therapy. The study will be conducted as a sub-study within the Hunter Outcome Survey (HOS). Hunter syndrome patients in the HOS who have previously received idursulfase as well as treatment-naive patients who will begin idursulfase treatment within 30 days of study enrollment will be included.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be considered eligible for enrollment:

* The patient is male and enrolled in the HOS (i.e., meets the entry criteria of a documented diagnosis of Hunter syndrome)
* The patient is ≥ 5 years-old
* The patient is on idursulfase treatment or scheduled to begin idursulfase treatment within 30 days of study enrollment
* The patient, patient's parent(s), or patient's legally authorized guardian must have voluntarily signed an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved informed consent form after all relevant aspects of the study have been explained and discussed with the patient, patient's parent(s), or patient's legally authorized guardian.

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for this study:

* The patient has received biologic/ERT products other than idursulfase, or other investigational product(s) for any reason within 30 days prior to study entry.
* The patient has a life expectancy of < 2 years
* The patient is unable to comply with the protocol, e.g., has a clinically relevant medical condition making implementation of the protocol difficult; has an uncooperative attitude; is unable to return for safety evaluations; or is otherwise unlikely to complete the study, as determined by the Investigator.

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Hunter syndrome
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2008-10-14 (Actual); Primary Completion 2013-02-08 (Actual); Study Completion 2013-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (6):
- United States (2):
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Children's Hospitals and Clinics of Minnesota, Division of Genetics, Minneapolis, Minnesota
- Hospital de Clinicas de Porto Alegre, Servico de Genetica Medica, Porto Alegre, Rio Grande do Sul, Brazil
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham
  - Great Ormond Street Hospital, London
  - Central Manchester University Hospitals, St. Mary's Hospital, Manchester

REFERENCES:
- [Result] Giugliani R, Harmatz P, Jones SA, Mendelsohn NJ, Vellodi A, Qiu Y, Hendriksz CJ, Vijayaraghavan S, Whiteman DA, Pano A. Evaluation of impact of anti-idursulfase antibodies during long-term idursulfase enzyme replacement therapy in mucopolysaccharidosis II patients. Mol Genet Metab Rep. 2017 Feb 21;12:2-7. doi: 10.1016/j.ymgmr.2017.01.014. eCollection 2017 Sep. PMID 28243577

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Elaprase® (0.5 mg/kg)
Started | 26
Completed | 15
Not Completed | 11
Not completed — Death | 2
Not completed — Other | 3
Not completed — Lost to Follow-up | 2
Not completed — Termination By Investigator | 3
Not completed — Withdrawal Of Consent | 1

BASELINE CHARACTERISTICS:
Arm/Group | Elaprase® (0.5 mg/kg)
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.82 (8.012)
Age, Customized [Count of Participants; unit: Participants]
  <12 years | 17
  ≥12 Years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 26
Region of Enrollment [Count of Participants; unit: Participants]
  BRAZIL | 6
  UNITED KINGDOM | 14
  UNITED STATES | 6

OUTCOME MEASURES:

1. Primary Outcome: Infusion-Related Adverse Event (IRAE) Rates Between IgG Anti-idursulfase Antibody Positive (Ab+) and Anti-idursulfase IgG Antibody Negative (Ab-) Patients
Description: The primary analysis of how presence of antibodies affected IRAE rates was performed based on a negative binomial regression model. This was done to account for potentially differential follow-up time between antibody groups.
Time Frame: Baseline to 109 Weeks
Population: The Safety Population was defined as all enrolled patients who received any portion of a dose of Elaprase.
Measure: Number; unit: IRAE/Week
Groups:
- Idursulfase (Elaprase) 0.5 mg/kg Weekly: Idursulfase: Patients will receive idursulfase as prescribed by their physician following locally approved prescribing information. Patients will not be provided idursulfase by Shire or the HOS.
Arm/Group | Idursulfase (Elaprase) 0.5 mg/kg Weekly
Number analyzed (Participants) | 26
IRAE/Week
  Ab+ (n =13) | 0.0121
  Ab- (n = 13) | 0.0042
  Ab+ (age adjusted)(n = 13) | 0.0055
  Ab- (age adjusted)(n = 13) | 0.0026
Statistical Analysis 1: Comparison: Idursulfase (Elaprase) 0.5 mg/kg Weekly; The groups compared are Ab+ vs Ab-; Test type: Superiority or Other; p = 0.1309, Negative Binomial Model; Relative Risk = 2.873, 95% CI 2-sided [0.731 to 11.296]
Statistical Analysis 2: Comparison: Idursulfase (Elaprase) 0.5 mg/kg Weekly; The groups compared are Ab+ (age adjusted) vs Ab- (age adjusted); Test type: Superiority or Other; p = 0.2718, Negative Binomial Model; Relative Risk = 2.082, 95% CI 2-sided [0.563 to 7.706]

2. Secondary Outcome: Change From Baseline in uGAG Levels to 109 Weeks
Description: Urine GAG
Time Frame: Baseline to 109 Weeks
Population: The Safety Population was defined as all enrolled patients who received any portion of a dose of Elaprase. The primary analysis of how presence of antibodies affected IRAE rates was performed based on a negative binomial regression model. This was done to account for potentially differential follow-up time between antibody groups.
Measure: Mean (Standard Deviation); unit: mcg/mg
Groups:
- Elaprase: Idursulfase 0.5 mg/kg Weekly Idursulfase: Patients will receive idursulfase as prescribed by their physician following locally approved prescribing information. Patients will not be provided idursulfase by Shire or the HOS.
Arm/Group | Elaprase
Number analyzed (Participants) | 15
mcg/mg | -74.07 (246.663)

ADVERSE EVENTS:
Arm/Group | Elaprase® (0.5 mg/kg)
Serious Adverse Events (participants affected / at risk) | 16/26
Other Adverse Events (participants affected / at risk) | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elaprase® (0.5 mg/kg) (N=26)
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Dental caries (Gastrointestinal disorders) | 1 (1)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1)
Hernia obstructive (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Central line infection (Infections and infestations) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Brain stem auditory evoked response (Investigations) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 2 (3)
Convulsion (Nervous system disorders) | 5 (6)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Neurological decompensation (Nervous system disorders) | 1 (1)
Syringomyelia (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic valve replacement (Surgical and medical procedures) | 1 (1)
Catheterisation venous (Surgical and medical procedures) | 1 (1)
Gastrostomy tube insertion (Surgical and medical procedures) | 1 (1)
Spinal operation (Surgical and medical procedures) | 1 (1)
Tonsillectomy (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elaprase® (0.5 mg/kg) (N=26)
Deafness (Ear and labyrinth disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 3 (9)
Eye pruritus (Eye disorders) | 2 (2)
Eye swelling (Eye disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 6 (8)
Diarrhoea (Gastrointestinal disorders) | 6 (11)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (13)
Adverse drug reaction (General disorders) | 2 (5)
Asthenia (General disorders) | 2 (2)
Catheter related complication (General disorders) | 3 (7)
Fatigue (General disorders) | 3 (3)
Gait disturbance (General disorders) | 2 (2)
Influenza like illness (General disorders) | 2 (2)
Infusion site extravasation (General disorders) | 2 (5)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 14 (43)
Seasonal allergy (Immune system disorders) | 2 (2)
Balanitis candida (Infections and infestations) | 2 (3)
Catheter site infection (Infections and infestations) | 2 (3)
Central line infection (Infections and infestations) | 2 (2)
Ear infection (Infections and infestations) | 9 (20)
Gastroenteritis (Infections and infestations) | 4 (4)
Influenza (Infections and infestations) | 4 (8)
Lower respiratory tract infection (Infections and infestations) | 9 (23)
Nasopharyngitis (Infections and infestations) | 3 (9)
Oral candidiasis (Infections and infestations) | 3 (5)
Otitis externa (Infections and infestations) | 4 (5)
Otitis media (Infections and infestations) | 3 (4)
Pharyngitis (Infections and infestations) | 2 (4)
Staphylococcal infection (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 12 (25)
Contusion (Injury, poisoning and procedural complications) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 9 (14)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Body temperature increased (Investigations) | 2 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (7)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2)
Convulsion (Nervous system disorders) | 6 (53)
Dizziness (Nervous system disorders) | 3 (4)
Grand mal convulsion (Nervous system disorders) | 2 (7)
Headache (Nervous system disorders) | 6 (31)
Paraesthesia (Nervous system disorders) | 2 (4)
Petit mal epilepsy (Nervous system disorders) | 5 (6)
Poor quality sleep (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (4)
Choking (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (25)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (9)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Skin chapped (Skin and subcutaneous tissue disorders) | 2 (2)
Central venous catheter removal (Surgical and medical procedures) | 2 (2)
Flushing (Vascular disorders) | 2 (5)
Hypertension (Vascular disorders) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤180 days from the time submitted to Shire for review. Shire does not prohibit publication, but can require the removal of confidential information (excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication.